CLINICAL TRIAL: NCT04034407
Title: Prospectively Randomized Controlled Trial on Damage Control Surgery for Perforated Diverticulitis With Generalized Peritonitis
Brief Title: Trial on Damage Control Surgery for Perforated Diverticulitis With Generalized Peritonitis
Acronym: Damage Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Version 1.03
Record Dates: First submitted 2019-07-22; First posted 2019-07-26 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Damage Control for Perforated Diverticulitis

STUDY DESIGN:
Intervention Model Description: 1:1 randomization to damage control surgery or control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Damage control surgery (Experimental): In the damage control surgery (DCS) group the surgeon was asked to perform rapid source control by stapling the perforated segment leaving blind ends or suturing the perforation site if possible, doing a thorough lavage of the abdominal cavity and placing an intra-abdominal negative pressure system avoiding the retraction of the abdominal wall with dynamic sutures as published. The second-look operation was scheduled for a time 24-48 hours after primary surgery that would be during regular working hours with a colorectal surgeon on hand to make the decision for either anastomosis or ostomy.
  Interventions: Procedure: Damage control surgery
- Control group (Active Comparator): In the conventional treatment group (Group C), the decision to reconstruct the colon or perform a Hartmann procedure was made by the surgeon during the emergency operation. After performing the anastomosis or the Hartmann procedure, patients with advanced peritonitis received an intraabdominal negative pressure system at the discretion of the operating surgeon.
  Interventions: Procedure: Damage control surgery

INTERVENTIONS:
Procedure: Damage control surgery — All patients with clinical and radiological suspicion of colonic perforation and generalized Peritonitis with indication for emergency surgery were included in the study.
  Randomisation was performed intraoperatively in all patients after the performing surgeon confirmed a colonic perforation with generalized peritonitis.

SUMMARY:
Damage control surgery (DCS) with abdominal negative pressure therap (NPT) and delayed anastomosis creation in patients with perforated diverticulitis and generalized peritonitis was established at our Institution in 2006 and has been published. This is the first prospectively controlled randomized study comparing DCS with conventional treatment (Group C).

DETAILED DESCRIPTION:
Inclusion criteria:

All patients with clinical and radiological suspicion of colonic perforation and generalized Peritonitis with indication for emergency surgery were included in the study.

Exclusion criteria:

* Covered perforation or peritonitis limited to one quadrant
* No colonic perforation (gastric perforation, appendicitis, ...)
* Malignancy as cause of perforation
* Age < 18 years
* Pregnancy
* Preoperative anal incontinence
* No patient consent

Primary endpoint:

Reconstructed bowel continuity at discharge and 6 months.

Secondary endpoint:

* Permanent stoma rate
* 30-day mortality rate
* Postoperative complications

Randomisation was performed intraoperatively in all patients after the performing surgeon confirmed a colonic perforation with generalized Peritonitis. All patients preoperatively granted their consent to participate in the study.

Surgical strategy:

In the damage control surgery (DCS) group the surgeon was asked to perform rapid source control by stapling the perforated segment leaving blind ends or suturing the perforation site if possible, doing a thorough lavage of the abdominal cavity and placing an intra-abdominal negative pressure system avoiding the retraction of the abdominal wall with dynamic sutures as published. The second-look operation was scheduled for a time 24-48 hours after primary surgery that would be during regular working hours with a colorectal surgeon on hand to make the decision for either anastomosis or ostomy. In the conventional treatment group (Group C), the decision to reconstruct the colon or perform a Hartmann procedure was made by the surgeon during the emergency operation. After performing the anastomosis or the Hartmann procedure, patients with advanced peritonitis received an intraabdominal negative pressure system at the discretion of the operating surgeon.

Data collection and statistics:

Data were collected by our study nurse, who visited the patients, and statistical calculations were performed with SPSS 20. Assuming a reconstruction rate of 80% in the study group and 50% in the conventional treatment group, we calculated that 70 patients would be needed to prove our hypothesis. Statistical calculation was performed with Chi-square for distribution of clinical data and stoma rate and the Mann-Whitney U test was used to compare numeric and nonparametric data. The study was approved by our local ethics committee (EC No.: UN5157).

ELIGIBILITY:
Inclusion Criteria:

* All patients with clinical and radiological suspicion of colonic perforation and generalized Peritonitis with indication for emergency surgery were included in the study and intraoperatively confirmed generalized peritonitis

Exclusion Criteria:

* Covered perforation or peritonitis limited to one quadrant
* No colonic perforation (gastric perforation, appendicitis, ...)
* Malignancy as cause of perforation
* Age < 18 years
* Pregnancy
* Preoperative anal incontinence
* No patient consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-10-14 (Actual); Primary Completion 2018-10-14 (Actual); Study Completion 2018-10-14 (Actual)

PRIMARY OUTCOMES:
Reconstructed bowel continuity | 4 weeks
  Patients leaving the hospital with complete bowel reconstruction.

SECONDARY OUTCOMES:
Reconstructed bowel continuity | 6 months
Permanent stoma rate | 1 year
  Patients with permanent colostomy.
Mortality rate | 30-days
Postoperative complications | 90-days
  Any complication during hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Reinhold Kafka-Ritsch, Dr., Principal Investigator — Innsbruck Medical University, Dept. of Visceral, Transplant and Thoracic Surgery

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kafka-Ritsch R, Birkfellner F, Perathoner A, Raab H, Nehoda H, Pratschke J, Zitt M. Damage control surgery with abdominal vacuum and delayed bowel reconstruction in patients with perforated diverticulitis Hinchey III/IV. J Gastrointest Surg. 2012 Oct;16(10):1915-22. doi: 10.1007/s11605-012-1977-4. Epub 2012 Jul 28. PMID 22843083
- [Background] Perathoner A, Klaus A, Muhlmann G, Oberwalder M, Margreiter R, Kafka-Ritsch R. Damage control with abdominal vacuum therapy (VAC) to manage perforated diverticulitis with advanced generalized peritonitis--a proof of concept. Int J Colorectal Dis. 2010 Jun;25(6):767-74. doi: 10.1007/s00384-010-0887-8. Epub 2010 Feb 11. PMID 20148255
- [Derived] Kafka-Ritsch R, Zitt M, Perathoner A, Gasser E, Kaufman C, Czipin S, Aigner F, Ofner D. Prospectively Randomized Controlled Trial on Damage Control Surgery for Perforated Diverticulitis with Generalized Peritonitis. World J Surg. 2020 Dec;44(12):4098-4105. doi: 10.1007/s00268-020-05762-1. Epub 2020 Sep 8. PMID 32901323
- See also: Clinical Trial Registry of the Tirol Kliniken GmbH — https://ctc.tirol-kliniken.at/page.cfm?vpath=oeffentliche&action=viewdetail&studie=6411